CLINICAL TRIAL: NCT02752256
Title: Quality and Effectiveness of Thrombolytic Care During Inter-hospital Transfer ("Drip-Ship") With Air Ambulance Services
Brief Title: Thrombolytic Care During Inter-hospital Transfer
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Brett A Faine, Clinical Pharmacy Specialist, University of Iowa
Other Study IDs: IRB:201507803
Record Dates: First submitted 2016-04-18; First posted 2016-04-26 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Stroke
Keywords: tissue plasminogen activator
MeSH Terms: conditions — Stroke | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intervention/Transfer: Patients who are transferred via air ambulance to a comprehensive stroke center
  Interventions: Drug: Tissue Plasminogen Activator
- Control: Patients presenting directly to the comprehensive stroke center
  Interventions: Drug: Tissue Plasminogen Activator

INTERVENTIONS:
Drug: Tissue Plasminogen Activator

SUMMARY:
Evaluation of ischemic stroke patients receiving tissue plasminogen activator (rtPA) during air ambulance transfer

DETAILED DESCRIPTION:
The purpose of our study is to evaluate the effect of air ambulance transport on patients presenting with an ischemic stroke and receive tissue plasminogen activator (rtPA). Primary outcome will be the evaluation of air ambulance transfer and if it leads to protocol violations or significant delays in therapy. Protocol violations include inaccurate dosing or preparation at the outside hospital, uncontrolled blood pressure before and during the flight, unnecessary medication administration before and during the flight and adverse events (intracranial bleeding, allergic reaction) associated with transfer process. Additional evaluation will include the effects of vibration of the air ambulance and its effects on the lytic activity of rtPA. rtPA is not supposed to be significantly agitated after it is prepared in solution and there is significant vibration and agitation during air ambulance transfer.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received tissue plasminogen activator for acute ischemic stroke
* presented directly to comprehensive stroke center or were transferred by our air ambulance service

Exclusion Criteria:

* Transferred by another air ambulance service or ground ambulance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All acute ischemic stroke patients who receive rtPA and transferred to our institution via our air ambulance service or present directly to our ED
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2015-10; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

REFERENCES:
- [Derived] Faine BA, Dayal S, Kumar R, Lentz SR, Leira EC. Helicopter "Drip and Ship" Flights Do Not Alter the Pharmacological Integrity of rtPA. J Stroke Cerebrovasc Dis. 2018 Oct;27(10):2720-2724. doi: 10.1016/j.jstrokecerebrovasdis.2018.05.049. Epub 2018 Jul 20. PMID 30037651

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention/Transfer: Patients who are transferred via air ambulance to a comprehensive stroke center
  Tissue Plasminogen Activator
- Control: Patients presenting directly to the comprehensive stroke center
  Tissue Plasminogen Activator
Period: Overall Study
Arm/Group | Intervention/Transfer | Control
Started | 35 | 41
Completed | 35 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention/Transfer | Control | Total
Number analyzed (Participants) | 35 | 41 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (14.3) | 65 (22.2) | 66 (18.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 20 | 35
  Male | 20 | 21 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 35 | 41 | 76
Region of Enrollment [Number; unit: participants]
  United States | 35 | 41 | 76
NIH Stroke Scale/Score (NIHSS) [Mean (Standard Deviation); unit: units on a scale] — Minimum 0 (good clinical outcome), Maximum 42 (poor clinical outcome)
  units on a scale | 8 (8) | 6 (5) | 7 (6)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a rtPA Protocol Violation
Description: Protocol violations can include any of the following recorded outcomes: inaccurate dosing or preparation at the outside hospital, uncontrolled blood pressure before and during the flight, unnecessary medication administration before and during the flight, intracranial bleeding, and angioedema
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention/Transfer | Control
Number analyzed (Participants) | 35 | 41
Participants | 7 | 0

2. Secondary Outcome: Average Time to rtPA
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Intervention/Transfer | Control
Number analyzed (Participants) | 35 | 41
Minutes | 74.5 (34.2) | 60 (31.2)

ADVERSE EVENTS:
Time Frame: In-hospital mortality, serious adverse events, adverse events up to 90 days
Arm/Group | Intervention/Transfer | Control
All-Cause Mortality (participants affected / at risk) | 2/35 | 1/41
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/41
Other Adverse Events (participants affected / at risk) | 0/35 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-11): https://cdn.clinicaltrials.gov/large-docs/56/NCT02752256/Prot_SAP_000.pdf